CLINICAL TRIAL: NCT03240783
Title: A Comparative Effectiveness Randomised Placebo Controlled Pilot Trial of the Management of Acute Lumbar Radicular Pain: Evaluate Route Versus Pharmacology of Intervention, and Feasibility in Public Hospital and Community Practice Settings.
Brief Title: A Comparative Effectiveness Randomised Placebo Controlled Pilot Trial of the Management of Acute Lumbar Radicular Pain
Acronym: SCIATICA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George Hospital, Australia (Other)
Collaborators: St George & Sutherland Medical Research Foundation (Unknown)
Responsible Party: Principal Investigator, Marissa Lassere, Principal Investigator, St George Hospital, Australia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: StGeorgeH
Record Dates: First submitted 2017-07-31; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Acute Sciatica
Keywords: CT-Fluoroscopic Selective Transforaminal Epidural Steroid; Oral Dexamethasone; Acute Lumbar Radiculopathy; Sciatic Neuropathy; Betamethasone injectable; Dexamethasone injectable; Acute Lumbar radicular pain; Randomized Controlled Trial (RCT); Comparative Effectiveness Controlled Trial
MeSH Terms: conditions — Sciatic Neuropathy | interventions — Betamethasone; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Randomised 1:1:1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care-provider (general-practitioner and/or specialist), investigator, and outcomes assessor are masked to the treatment arms. All personnel except the radiologist delivering the procedure and the investigator responsible for randomisation will be masked to the randomisation arm. The participant, study personnel, other investigators, participant's treating physician and study analyst will be blind to the results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm 1 (Experimental): Betamethasone OR Dexamethasone Injectable CT - fluoroscopic guided transforaminal lumbar epidural steroid
  Interventions: Drug: Betamethasone OR Dexamethasone Injectable; Other: Sham Injection and/or oral placebo
- Arm 2 (Experimental): Normal Saline Flush, 0.9% Injectable Solution CT - fluoroscopic guided transforaminal lumbar epidural normal saline
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution; Other: Sham Injection and/or oral placebo
- Arm 3 (Experimental): Dexamethasone Oral Tablet:
  Oral dexamethasone 15 day tapered dosing is as follows: (i) days 1-5, 4 mg morning and evening, (ii) days 6-10, 2 mg morning and evening, and (iii) days 11-15, 1mg morning and evening.
  Interventions: Drug: Dexamethasone Oral Tablet; Other: Sham Injection and/or oral placebo
- Arm 4 (Other): Sham Injection and/or oral placebo: CT/fluoroscopic guided (parameters set to zero) transforaminal lumbar sham (needle placement down to muscle and no injection of any fluid) AND placebo oral tablets taper.
  Interventions: Other: Sham Injection and/or oral placebo

INTERVENTIONS:
Drug: Betamethasone OR Dexamethasone Injectable — Procedural agents. The steroid and local anaesthetic preparation will be standardized to replicate current radiology interventional practices that use either particulate or non-particulate steroids. Betamethasone Sodium Phosphate/Acetate 5.7 mg/ml Injectable is a particulate corticosteroid and is used with the local anaesthetic bupivacaine 0.5% (1ml). Dexamethasone 4mg (1ml) is a non-particulate corticosteroid and is used with the local anaesthetic lignocaine 1% (1ml).
  Other Names: celestone chondrase 5.7 mg/ml injectable suspension
  Arms: Arm 1
Drug: Normal Saline Flush, 0.9% Injectable Solution — Procedural agents. The local anaesthetic preparation used with the Normal Saline Flush, 0.9% Injectable Solution, will be standardized to replicate current radiology interventional practices: either local anaesthetic bupivacaine 0.5% (1ml) or local anaesthetic lignocaine 1% (1ml).
  Other Names: There is no other name.
  Arms: Arm 2
Drug: Dexamethasone Oral Tablet — Dexamethasone Oral Tablet: 15 day taper dosing is: days 1-5 8mg (4mg bd) , days 6-10 4 mg (2mg bd), and days 11-15 2 mg (1mg bd). The dexamethasone is over-encapsulated in a gelatine capsule that is identical to the placebo capsule in appearance.
  Other Names: Dexmethsone
  Arms: Arm 3
Other: Sham Injection and/or oral placebo — The sham Injection procedure is needle placement down to muscle at the designated spinal level and no injection of any fluid. The oral placebo is a gelatine capsule packed with filler.
  Other Names: There is no other name

SUMMARY:
Aim: In subjects with acute sciatica (≤ 4 weeks duration), this is a pilot comparative effectiveness study to evaluate feasibility and to determine final sample size for a future adequately powered randomised controlled trial of (i) CT-guided transforaminal lumbosacral epidural steroid injection, and (ii) oral dexamethasone, in a masked (blinded), randomised, sham injection and oral placebo controlled trial.

Study Design: 60 patients with acute sciatica will randomised 1:1:1:1 to receive either (i) epidural steroid injection & oral placebo, (ii) epidural normal saline injection & oral placebo, (iii) oral dexamethasone & IM sham-injection, (iv) IM sham-injection & oral placebo.

Outcomes: The primary outcome is reduction of disability at 3 weeks using the Oswestry Disability Index. Secondary outcomes include reduction of disability at 6 and 48 weeks.

DETAILED DESCRIPTION:
Acute sciatica, a major cause of pain and disability, is a common presentation to medical practices and hospitals. Up to 25% of patients do not recover after 12 months. Sciatica refers to radicular pain and radiculopathy from lumbosacral nerve root pathology caused by lumbosacral disc herniation and degenerative lumbosacral spondylosis involving the L2/3 to L5/S1 intervertebral discs and foramina. Selective transforaminal epidural steroid injection and systemic steroids are therapeutic options in patients who do not improve with conservative management. However, there is limited evidence of effectiveness of these treatments in acute sciatica.

This pilot study is designed to evaluate the following feasibility and study conduct issues: type and standardization of interventions and associated sham and placebo control, appropriateness of inclusion and exclusion criteria, rate of recruitment, study conduct including randomisation allocation concealment, successful masking, wait time for delivery of services (allied health, diagnostic imaging, and procedures), and ensuring efficient, appropriate and safe study conduct for recruitment from emergency departments, hospital inpatients, general practitioners and specialists in the community, and radiology departments in hospital and community practices. Study logistics will differ across these settings, and processes to ensure standardization will be evaluated. Other issues explored include co-therapy with analgesics, NSAIDS, pregabalin, physical and manual therapies, and the timing of rescue therapy, including neurosurgery. It is our experience with previous RCTs that piloting all facets and procedures is essential for the successful conduct of a RCT.

Furthermore, results of the categorical and continuous primary and secondary outcomes from this pilot RCT will be used to calculate the sample size of an adequately powered RCT to determine which treatments currently used in the management of acute sciatica/lumbosacral radiculopathy of less than 4 weeks duration, is the most effective in reducing pain and disability in the short-term and prevent progression to persistent or recurrent sciatica/lumbosacral radiculopathy in the long term.

Study Design: 60 patients with acute sciatica will randomised 1:1:1:1

Arm 1: CT - fluoroscopic guided transforaminal lumbar epidural steroid (1 ml) mixed with local anaesthetic (1 ml) (Active Intervention) AND oral placebo taper (Placebo Control) Note: The injectable steroid and local anaesthetic preparation is standardized to replicate current practice: EITHER (i) betamethasone injectable 5.7 (1ml), a particulate corticosteroid with the local anaesthetic bupivacaine 0.5% (1ml) OR (ii) dexamethasone injectable 4mg (1ml) a non-particulate corticosteroid with local anaesthetic lignocaine 1% (1ml).

Arm 2: CT - fluoroscopic guided transforaminal lumbar epidural normal saline (1 ml) mixed with local anaesthetic (1ml) (Active Intervention controlling for pharmacology) AND oral placebo taper (Placebo Control) Note: The Normal Saline is a Normal Saline flush 0.9% injectable solution. The local anaesthetic preparation is standardized to replicate current practice: EITHER (i) bupivacaine 0.5% (1ml) OR (ii) lignocaine 1% (1ml).

Arm 3: Oral dexamethasone taper (Active Intervention) AND sham injection (Sham Control) Oral dexamethasone taper is a 15 day tapered dosing: (i) days 1-5, dexamethasone 4 mg morning and evening, (ii) days 6-10, dexamethasone 2 mg morning and evening, and (iii) days 11-15, dexamethasone 1mg morning and evening. The dexamethasone gelatine capsule is identical to the placebo capsule in appearance. The sham injection is CT/fluoroscopic guided (with parameters set to zero) lumbar sham injection. The needle placement is down to muscle layer but NOT into the epidural space, and there is no injection of any fluid.

Arm 4: Sham injection (Sham Control) AND oral placebo taper (Placebo Control) The sham injection is CT/fluoroscopic guided (with parameters set to zero) lumbar sham injection. The needle placement is down to muscle layer but NOT into the epidural space, and there is no injection of any fluid. The oral placebo is a gelatine capsule with filler. It is identical to the dexamethasone capsule in appearance.

Participants: If eligibility criteria are met then participants will be invited to participate in the RCT. If the participant agrees, then the participant proceeds down study pathway. A log of all potential participants who are referred and screened and who either decline to participate in the RCT or deemed ineligible by the eligibility criteria will be kept. This will ascertain the representativeness of those who consent to be randomized, consistent with CONSORT guidelines. Data collected in the refusal/reject log will include age, gender, reason(s) for ineligibility or refusal, and, if available, pain/disability score and treatment.

Outcomes: The primary outcome is reduction of disability at 3 weeks using the condition-specific Oswestry Disability Index (ODI). Secondary outcomes include reduction of disability at 6 and 48 weeks on (ODI), Numerical Rating Scale (NRS) for leg pain and for back pain respectively, measures of generic function/disability and quality of life (SF-36, EQ-5D), length of hospital stay, medication co-therapy use (simple analgesics, opiate analgesics, pregabalin, and NSAIDs), need for rescue procedures or surgery, time to return to work (if applicable), compliance with treatment, masking success, measures of study conduct and efficiency, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Leg pain of any description with clinical findings consistent with single level radiculopathy
* Minimum symptom duration > 72hrs
* Maximum symptom duration < 3 weeks to ensure symptom duration at randomisation is ≤ 4 weeks
* No previous episode of same level radicular pain in the previous 6 months
* Pain intensity at >30 on the Oswestry Disability Index (ODI)
* Imaging (MRI and/or CT) indicating herniated disc or foraminal stenosis or both, concordant with the level indicated by history and physical examination

Exclusion Criteria:

* Previous transforaminal epidural steroids at any level in the last 12 months
* Previous oral steroids in the last 12 months
* Any lumbar surgery at same level, or above or below the level at any time
* Previous lumbar surgery at any other level to that in (iii) within the last 12 months
* Pregnancy, or lactation/breastfeeding
* Direct indication for neurosurgery (e.g. cauda equina syndrome, or progressive motor loss i.e. less than or equal to 3/5 power)
* Inability to read or understand English
* Any serious medical or psychiatric condition that may interfere with participation or outcome assessment such as: need for uninterrupted anti-coagulation, spinal fracture, active infection or metastatic disease suspected, active cancer, poorly controlled diabetes, or patients with diabetes on any insulin, uncontrolled hypertension (systolic blood pressure >180 or diastolic blood pressure >110 within 30 days of randomization date), active peptic ulcer disease, history of intolerance to steroid therapy, previous or current psychiatric history of bipolar disease, or secondary gain such as anticipated or ongoing legal proceedings, history of substance abuse

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-08 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) version 2.0 | 3 weeks
  ODI is a functional status measure specifically developed for disorders of the spine

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) version 2.0 | 6 weeks
  ODI is a functional status measure specifically developed for disorders of the spine
Oswestry Disability Index (ODI) version 2.0 | 12 weeks
  ODI is a functional status measure specifically developed for disorders of the spine
Oswestry Disability Index (ODI) version 2.0 | 48 weeks
  ODI is a functional status measure specifically developed for disorders of the spine
Numerical Rating Scale (NRS) for leg pain | 3 weeks
  The NRS is a validated 11 point scale
Numerical Rating Scale (NRS) for leg pain | 6 weeks
  The NRS is a validated 11 point scale
Numerical Rating Scale (NRS) for leg pain | 12 weeks
  The NRS is a validated 11 point scale
Numerical Rating Scale (NRS) for leg pain | 48 weeks
  The NRS is a validated 11 point scale

OTHER OUTCOMES:
Short-Form 36 (SF-36) questionnaire | 1, 3, 6, 12, and 48 weeks
  health related quality of life
EuroQol 5D | 1, 3, 6, 12, and 48 weeks
  quality-adjusted-life-year using QALYs
Work and health utilisation | 1, 3, 6, 12, and 48 weeks
  days missed from paid employment (if applicable) because of sciatica, use of health services such as doctor, other health-care provider related visits (acupuncture, chiropractic), repeat epidurals and surgical procedures
Adverse events | 1, 3, 6, 12, and 48 weeks
  These will include steroid adverse effects (blood pressure, blood glucose, changes in mood and sleep) and procedural adverse effects (headaches, bleeding) and information about additional procedures, surgery and hospitalisations.
Masking success | Day 0, Day 1, Weeks 1, 3, 6 and 12
  Whether participants, outcome assessors and investigators were successfully masked to study randomised arms

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Lassere, MBBS PhD, Principal Investigator — St George Hospital SESLHD
Locations (1):
- St George Hospital, Kogarah, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lassere MN, Johnson KR, Thom J, Pickard G, Smerdely P. Protocol of the randomised placebo controlled pilot trial of the management of acute sciatica (SCIATICA): a feasibility study. BMJ Open. 2018 Jul 5;8(7):e020435. doi: 10.1136/bmjopen-2017-020435. PMID 29980542